CLINICAL TRIAL: NCT01785641
Title: Single Versus Combined Antibiotic Therapy for Bacterial Peritonitis in Continuous Ambulatory Peritoneal Dialysis Patients
Brief Title: Single Versus Combined Antibiotic Therapy for Bacterial Peritonitis in CAPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RA56/006
Record Dates: First submitted 2013-01-30; First posted 2013-02-07 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2013-02

CONDITIONS: Peritonitis
Keywords: peritoneal dialysis; peritonitis
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ceftazidime+ciprofloxacin (Experimental): 2 synergistic antibiotics(ceftazidime IP and ciprofloxacin po for gram negative bacterial peritonitis)
  Interventions: Drug: ceftazidime+ciprofloxacin
- ceftazidime monotherapy (Active Comparator): ceftazidime IP for gram negative bacterial peritonitis
  Interventions: Drug: ceftazidime monotherapy
- cefazolin+gentamicin (Experimental): cefazolin IP and gentamicin IP for gram positive bacterial peritonitis
  Interventions: Drug: cefazolin+gentamicin
- cefazolin monotherapy (Active Comparator): cefazolin IP for gram positive bacterial peritonitis
  Interventions: Drug: cefazolin monotherapy

INTERVENTIONS:
Drug: ceftazidime+ciprofloxacin — 2 synergistic antibiotics: ceftazidime IP + ciprofloxacin po for gram negative bacterial peritonitis
  Other Names: combined antibiotic therapy
  Arms: ceftazidime+ciprofloxacin
Drug: ceftazidime monotherapy — ceftazidime IP for gram negative bacterial peritonitis
  Other Names: monotherapy
  Arms: ceftazidime monotherapy
Drug: cefazolin+gentamicin — cefazolin IP + gentamicin IP for gram positive bacterial peritonitis
  Other Names: combined antibiotic therapy
  Arms: cefazolin+gentamicin
Drug: cefazolin monotherapy — cefazolin IP for gram positive bacterial peritonitis
  Other Names: monotherapy
  Arms: cefazolin monotherapy

SUMMARY:
To compare the efficacy of single versus combined antibiotic therapy for bacterial peritonitis in CAPD patients.

DETAILED DESCRIPTION:
To compare relapse and recurrent rate of peritonitis between single and combined antibiotic regimens for bacterial peritonitis in CAPD patients.

ELIGIBILITY:
Inclusion Criteria:

* age >/= 18 years old
* ESRD patients on continuous ambulatory peritoneal dialysis more than 4 weeks
* presence of symptom or sign of peritonitis
* presence of WBC >100cell/mm3 with PMN >50% in peritoneal dialysate or gram stain positive for gram positive or gram negative bacteria

Exclusion Criteria:

* presence of polymicrobial organism, non-fermentative gram negative organism, fungus, mycobacteria in peritoneal fluid or culture-negative
* peritonitis from the organisms that required combined antibiotic therapy according to ISPD guideline 2010
* hospital-acquired peritonitis
* presence of catheter-related infection
* history of peritonitis within 4 weeks
* currently taking antibiotic
* allergic to the antibiotic that used in the study(penicillin or cephalosporin or quinolone or aminoglycoside)

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
relapse or recurrent rate | within 4 weeks after peritonitis treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nalinee Saiprasertkit, MD., Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn university, Bangkok, Thailand